CLINICAL TRIAL: NCT03983512
Title: The PULSTA Transcatheter Pulmonary Valve (TPV) Pre-Approval Study
Brief Title: PULSTA Transcatheter Pulmonary Valve Pre-Approval Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taewoong Medical Co., Ltd. (Industry)
Collaborators: Avania (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TWTPV-E1001
Record Dates: First submitted 2019-06-07; First posted 2019-06-12 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Heart Diseases; Pulmonary Valve Regurgitation; Pulmonary Valve Stenosis; Tetralogy of Fallot
MeSH Terms: conditions — Heart Diseases; Pulmonary Valve Insufficiency; Pulmonary Valve Stenosis; Tetralogy of Fallot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PULSTA TPV (Experimental): PULSTA Transcatheter Pulmonary Valve (TPV) System
  Interventions: Device: PULSTA TPV System

INTERVENTIONS:
Device: PULSTA TPV System — PULSTA transcatheter pulmonary valve replacement.

SUMMARY:
The purpose of the study is to evaluate the safety and effectiveness of the PULSTA Transcatheter Pulmonary Valve (TPV) System for the treatment of congenital or acquired pulmonary valve stenosis and/or regurgitation who require pulmonary valve replacement.

DETAILED DESCRIPTION:
The PULSTA TPV is a self-expandable valve with flared-ends to adapt to the larger native right ventricular outflow tract (RVOT) and is using a relatively low profile delivery catheter from knitted nitinol wire backbone and trileaflets made from treated porcine pericardial tissue, and a delivery system, which provides access to the right ventricular outflow tract through blood vessels. Consecutive subject data should be collected at discharge, 1, 6 months, and 1-5 years post PULSTA TPV implantation.

ELIGIBILITY:
Inclusion Criteria:

* Body weight greater than or equal to 30 kilograms
* Pulmonary regurgitation moderate or severe pulmonary regurgitation or pulmonary valve stenosis with mean gradient >35mmHg by echocardiography
* Main pulmonary artery trunk of ≥16 mm and ≤30 mm
* Patients willing to provide written informed consent and comply with follow-up evaluations.

Exclusion Criteria:

* Females of child-bearing potential who are unable to take adequate contraceptive precautions, are known to be pregnant, or are currently breastfeeding an infant up until 6 months after TPV implantation
* Pre-existing mechanical valve in pulmonary position or require concomitant repair of other cardiac valves
* Obstruction of the central veins to be approached for the TPV implantation
* Coronary artery compression confirmed by angiography
* A known severe allergy to Nickel
* A known hypersensitivity to any anticoagulation therapy, contrast agent or a hemorrhagic disease
* Suspected active infectious disease (e.g. endocarditis, meningitis)
* Life expectancy of less than 6 months

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2019-10-07 (Actual); Primary Completion 2022-09-21 (Actual); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Procedural/Device related serious adverse events at 6 months | 6 months
Hemodynamic functional improvement at 6 months | 6 months
  Hemodynamic functional improvement is a composite of mean RVOT gradient ≤30 mmHg by continuous wave Doppler and a pulmonary regurgitant fraction <20% by cardiac magnetic resonance (MR)

SECONDARY OUTCOMES:
Procedural Success | 7 days
  Procedural success is defined as the TPV implant within desired position, Right ventricle-Pulmonary artery (RV-PA) peak systolic pressure gradient <35mmHg by catheter, less mild pulmonary regurgitation by angiography, and freedom from explantation of the TPV at 24 hours post-implant.
Hemodynamic Function | 5 years
  Hemodynamic function will be assessed including peak RVOT pressure gradient, mean RVOT pressure gradient, right ventricle (RV) end-diastolic volume index by echocardiography or cardiac MR.
Pulmonary Regurgitant Fraction | 6months
  Pulmonary regurgitant fraction (PRF) will be assessed via cardiac MRI at 6 months after the PULSTA TPV implantation.
Severity of Pulmonary Regurgitation | 5 years
  Severity of pulmonary regurgitation will be assessed via Doppler echocardiography.
NYHA functional classification | 5 years
  Clinical outcome will be assessed as per the New York Heart Association (NYHA) functional classification t all follow-up visits and will be compared to baseline values.
Catheter reintervention on TPV | 5 years
  Catheter re-intervention on PULSTA TPV is defined as any interventional catheter procedure (e.g. balloon angioplasty) that alters or adjusts, or replaces a previously implanted PULSTA TPV during a 5-year follow-up period, and the frequency will be evaluated.
Reoperation | 5 years
  Reoperation is defined as open surgery that alters or adjusts, or replaces a previously implanted PULSTA TPV during a 5-year follow-up period, and the frequency will be evaluated.
Procedural / Device related serious adverse events | 5 years
Death (All cause / procedural/device-related) | 5 years
Other adverse events | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Mario Carminati, PhD. MD., Study Chair — Policlinico San Donato; Stanimir Georgiev, PhD. MD., Principal Investigator — Deutsches Herzzentrum Munchen; Jose Luis Zunzunegui, PhD. MD., Principal Investigator — Gregorio Marañon hospital; Federico Gutierrez Larraya, PhD. MD., Principal Investigator — Hospital Universitario La Paz; Ender Odemis, PhD. MD., Principal Investigator — Koc University Hospital; Ahmet Çelebi, PhD. MD., Principal Investigator — Siyami Ersek Hospital; Gregor Krings, PhD. MD., Principal Investigator — Utrecht University Wilhelmina; Thomas Krasemann, PhD. MD., Principal Investigator — Erasmus Medical Center; Gi Beom Kim, PhD. MD., Principal Investigator — Seoul National University Hospital; Jae Young Choi, PhD. MD., Principal Investigator — Severance Hospital; Seong Ho Kim, PhD. MD., Principal Investigator — Sejong General Hospital
Locations (11):
- Deutsches Herzzentrum Munchen, München, München, Germany
- Policlinico San Donato, Milan, San Donato Milanese, Italy
- Netherlands (2):
  - Utrecht University Wilhelmina, Utrecht, Utrecht
  - Erasmus Medical Center, Rotterdam, Wytemaweg
- South Korea (3):
  - Seoul National University Hospital, Seoul, Haehak-ro Jongno-gu
  - Sejong General Hospital, Bucheon-si, Hohyun-ro, Sosa-gu
  - Severance Hospital, Seoul, Yonsei-ro, Seodaemun-gu
- Spain (2):
  - Gregorio Marañon hospital, Madrid, Madrid
  - University Hospital La Paz, Madrid, Madrid
- Turkey (Türkiye) (2):
  - Koc University Hospital, Istanbul, Topkapı, Zetinburnu/İstanbul
  - Siyami Ersek Hospital, Istanbul, Üsküdar/İstanbul

IPD SHARING:
Plan to Share IPD: No